CLINICAL TRIAL: NCT05899322
Title: Adaptation and Translation of the Primary Care Intervention for PTSD for Spanish Speaking Adolescents and Families
Brief Title: Adaptation of the PCIP for Spanish Speaking Adolescents and Families
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Begun collaborating with a new community partner and will submit a new study with that partner.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lauren Ng, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #22-001744
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Post-Traumatic Stress Disorder in Adolescence; Post Traumatic Stress Disorder
Keywords: Primary Care; PTSD; Post Traumatic Stress Disorder; Randomized Pilot Feasibility Trial; Spanish speaking adaptation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Mixed methods (qualitative and quantitative) randomized pilot feasibility trial (n=10 to treatment and 10 to waitlist control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Care Intervention for PTSD (PCIP) Spanish Speaking Adolescents and Families (Experimental): This arm will receive the culturally adapted and translated PCIP intervention lasting from 1-3 weeks, and will complete baseline, post treatment, and 1-month follow up assessments.
  Interventions: Behavioral: Primary Care Intervention for PTSD Spanish Speaking Adolescents
- Waitlist Treatment as Usual (Active Comparator): Receive standard care treatment and will complete baseline, post treatment, and 1-month follow up assessments, and are offered translated and adapted PCIP treatment after conclusion of the study.
  Interventions: Behavioral: Waitlist Treatment as Usual

INTERVENTIONS:
Behavioral: Primary Care Intervention for PTSD Spanish Speaking Adolescents — This treatment ranges from 1-3 sessions which last 30-50 minutes per session. The first session will cover psychoeducation about PTSD symptoms in children that can be delivered to the adolescent with optional parent involvement. The first session will also teach the adolescent a breathing technique to combat the physiological impact of PTSD in children. The subsequent sessions will be tailored to meet the needs of the adolescent's most distressing PTSD symptom cluster including hyper arousal, negative changes in cognition and mood, avoidance, re-experiencing. Each session contains coping skills that address the adolescent's symptoms. This treatment will be delivered via telehealth and all materials have been developed in both Spanish and English.
  Arms: Primary Care Intervention for PTSD (PCIP) Spanish Speaking Adolescents and Families
Behavioral: Waitlist Treatment as Usual — Will receive treatment as usual at local clinic and are provided information on free or low cost mental health care referrals in the Los Angeles Area.
  Arms: Waitlist Treatment as Usual

SUMMARY:
This study will implement a brief Post-traumatic Stress Disorder (PTSD) intervention for children, the Primary Care Intervention for PTSD (PCIP) delivered through telehealth (computer or smart phone delivery), to 10 Spanish speaking youth and their families.

Mixed methods (qualitative and quantitative) randomized pilot feasibility trial (n=10 to treatment and 10 to waitlist control) to refine the intervention, study procedures, and explore effectiveness.

Following RE-AIM guidelines, the investigators will assess:

Reach: patient participation in intervention delivery (out of all those asked to participate) and retention rate (out of all those who consented to participate and completed at least two intervention sessions) Adoption: patients and their parents/guardians will complete screening and intervention satisfaction ratings.

To understand patient experiences with the intervention and to identify and explain positive or negative treatment mechanisms or effects, the investigators will conduct post-intervention semi-structured interviews with the participating patients, their parents/guardians, and with providers.

This treatment ranges from 1-3 sessions which last 30-50 minutes per session. The first session will cover psychoeducation about PTSD symptoms in children that can be delivered to the parent or both the parent and child. The first session will also teach the parent and child a breathing technique to combat the physiological impact of PTSD in children. The subsequent sessions will be tailored to meet the needs of the child's most distressing PTSD symptom cluster including hyper arousal, negative changes in cognition and mood, avoidance, re-experiencing. Each session contains coping skills that the parent and child can learn together. There is also material for parents to address behavior problems in youth. This treatment will be delivered via telehealth.

All treatment materials have been developed in both Spanish and English.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to the SHARK Program
* Patients must be at least 12 years old
* Screened for probable PTSD on Brief UCLA Reaction Index, or at provider discretion of clinical relevancy.
* If patient is under 18 years old, the patient's legal guardian is able and willing to provide informed consent for the patient to participate in the study in English or Spanish;
* Patient is able to complete study activities in English or Spanish.

Exclusion Criteria:

* Suicidal ideation with a plan within the last two weeks or a suicide attempt within the past 30 days;
* Patient is over the age of 22

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-12 (Estimated); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Knowledge | Day 0 baseline, 1 month follow-up
  Changes in levels of PTSD Knowledge measured by the PTSD Knowledge Test (0-14, higher scores indicating more PTSD knowledge)
Change in Self-Reported Arousal | Day 0 baseline, 1 month follow-up
  Changes in PTSD related arousal levels measured by the Self-Assessment Manikin (SAM; 0-24, higher scores indicating higher arousal)
Intervention Acceptability | post treatment, average 1 month after enrollment
  Qualitative interviews will include questions regarding acceptability of treatment including treatment via telehealth and barriers to treatment.
Intervention Engagement | post treatment, average 1 month after enrollment
  Data will be collected regarding participant completion of therapy, no show rates, and attendance.
Intervention Implementation | post treatment, average 1 month after enrollment
  Study therapists will complete qualitative interviews regarding intervention delivery feasibility and study protocols.

SECONDARY OUTCOMES:
Change in PTSD Symptoms | Day 0 baseline, 1 month follow-up
  Changes in PTSD related symptoms measured by the UCLA Child/Adolescent PTSD Reaction Index for DSM-5 Brief Screen (total 0-44; Higher scores indicate higher likelihood of PTSD and symptom-related distress and impairment
Change in Trauma Symptoms | Day 0 baseline, 1 month follow-up
  Changes in trauma related symptoms measured by The Child PTSD Symptom Scale (CPSS-5-SR) Self Report (total 0-80, Higher scores indicated greater symptom severity).
Change in Depression Symptoms | Day 0 baseline, 1 month follow-up
  Changes in depression symptoms measured by the Patient Health Questionnaire (PHQ-9;0-27; Higher scores indicate higher symptoms and likelihood of depression)
Change in Anxiety Symptoms | Day 0 baseline, 1 month follow-up
  Changes in anxiety symptoms measured by the Revised Children's Anxiety and Depression Scale (RCADS) Self Report (total 0-141, Higher scores indicating higher symptom severity).
Change in Functional Impairment | Day 0 baseline, 1 month follow-up
  Changes in functional impairment measured by The Columbia Impairment Scale (C.I.S.; 0-52, Higher scores indicate greater impairment).
Change in Substance Use | Day 0 baseline, 1 month follow-up
  Changes in substance use and misuse measured by CRAFFT Adolescent Substance Use Screen (0-9, Higher scores indicate higher risk for substance misuse).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Ng, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No